CLINICAL TRIAL: NCT03519685
Title: UCSF College Health Study: A Cluster Randomized Trial on Contraceptive Training and Education at Community Colleges
Brief Title: UCSF College Health Study on Contraceptive Training and Education at Community Colleges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A125604
Record Dates: First submitted 2018-03-21; First posted 2018-05-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Contraception
Keywords: Contraception; Hormonal contraception; Long-acting reversible contraception; Condoms; Emergency contraception; Family planning services
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contraceptive Training and Education (Experimental): Colleges assigned to this arm receive a one-day UCSF Continuing Medical Education (CME # MMC18087) accredited training on contraceptives and technical assistance. The training is for staff at the student health center and local health centers where they refer for contraceptive services. Students attending colleges assigned to this arm receive education about contraceptive methods and how to access services.
  Interventions: Behavioral: Contraceptive Training and Education
- Nutrition Education (Placebo Comparator): Students attending colleges assigned to this arm receive nutrition education about the impacts of sugar on health.
  Interventions: Behavioral: Placebo Nutrition Education

INTERVENTIONS:
Behavioral: Contraceptive Training and Education — Staff at the student health center and local health centers where they refer for contraceptive services will receive a CME-accredited education and training session and technical assistance. The one-day session emphasizes evidence-based and patient-centered contraceptive counseling and provision. Students attending colleges assigned to the intervention arm will receive materials and resources designed to educate young people about contraceptive methods and where to access services.
  Arms: Contraceptive Training and Education
Behavioral: Placebo Nutrition Education — Students attending colleges assigned to the nutrition education arm will receive materials and resources designed to educate young people about the impacts of sugar on health.
  Arms: Nutrition Education

SUMMARY:
The purpose of this study is to measure whether a training and education intervention for clinic staff and young women aged 18-25 on contraceptive methods, including intrauterine devices (IUDs) and the implant, will result in greater contraceptive knowledge and access among students in community colleges.

DETAILED DESCRIPTION:
In the US, young women aged 18-25 years have limited knowledge of contraception or pregnancy risks and often experience challenges in accessing reproductive health care. They have little familiarity with the full range of contraceptives, particularly long-acting reversible contraception (LARC) including the IUD and implant. This campus-level, multiple component intervention provides evidence-based contraceptive training and education to clinic staff and students in this age group attending community colleges in California and Texas.

ELIGIBILITY:
Inclusion Criteria:

This study involves two groups of human subjects: students at 28 community colleges and staff at the student health center and referral clinics.

Students must be:

* Female;
* Age 18-25;
* Speaks English;
* Sexually active (vaginal sex with a male partner) in the last year;
* Not currently pregnant;
* Does not want to become pregnant in the next 12 months;
* At risk of pregnancy (including not sterilized);
* Enrolled in the current term at the participating community college;
* First-time college students, meaning no college enrollment prior to the current academic year; and
* Willing to be contacted by email and telephone over the next 12 months.

Clinic staff must:

* Be employed by a participating clinic; and
* Offer clinical care, counseling or education for contraception at the clinic.

For colleges to be eligible to be study sites, they must:

* Be an accredited community college;
* Not share health center staff with a participating college site;
* Have no active LARC intervention; and
* Enroll students ages 18-25 years.

Exclusion Criteria:

* Students and clinic staff will be excluded if they do not meet the inclusion criteria.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2086 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change in student knowledge of full range of contraceptive methods (questionnaire) | Baseline, immediate post educational intervention session
  The outcome is measured by whether student knows of reversible methods including male condom, female condom, oral contraceptive pill, transdermal patch, vaginal ring, Depo-provera injectable, intrauterine device, subdermal implant, and emergency contraception.

SECONDARY OUTCOMES:
Change in student access to contraceptive services over 12 months, measured as whether student knows of or visited health services for contraceptives (questionnaire) | Baseline, 12 months
Change in willingness to use long-acting reversible contraception (LARC) (questionnaire) | Baseline, immediate post educational intervention session
Change in LARC use over 12 months (questionnaire) | Baseline, 12 months
Dual condom use at last sex, measured by student report of condom use together with another method of birth control at last vaginal sex (questionnaire) | Baseline, 6 months, 12 months

OTHER OUTCOMES:
Unintended pregnancy incidence | 12 months
  The researchers will measure pregnancy through questionnaires and urine pregnancy tests.
Certificate or degree completion (ordinal outcome including categories for on-time progression for graduation, delayed progression or dropout), measured by student report (questionnaire) | 12 months
Change in receipt of public assistance (questionnaire) | Baseline, 12 months
Likelihood of finding good job after college measured by questionnaire item asking student if she thinks she will find a good job after college (measured with Likert scale: very likely, likely, unlikely, very unlikely) | 12 months
Change in provider LARC practices (questionnaire) | Baseline, 12 months
Sub-analyses for change in student knowledge of full range of contraceptive methods (questionnaire) | Baseline, immediate post educational intervention session, 6 months
  The outcome is measured by whether student knows of reversible methods including male condom, female condom, oral contraceptive pill, transdermal patch, vaginal ring, Depo-provera injectable, intrauterine device, subdermal implant, and emergency contraception. The researchers will assess the outcome of student contraceptive knowledge by sociodemographic factors (age, race/ethnicity, parental education, health insurance, receipt of public assistance) and reproductive characteristics (parity, pregnancy intentions, male partner, prior contraceptive use).
Sub-analyses for change in student access to contraceptive services over 12 months, measured as whether student knew of or visited health services for contraceptives (questionnaire) | Baseline, 12 months
  The researchers will assess the outcome of contraceptive access by sociodemographic factors (age, race/ethnicity, parental education, health insurance, receipt of public assistance) and reproductive characteristics (parity, pregnancy intentions, male partner, prior contraceptive use). The researchers will also test interaction of the intervention with race/ethnicity, parental education, and health insurance.
Sub-analyses for changes in LARC use over 12 months, measured by whether student is using an IUD or implant (questionnaire) | Baseline, 12 months
  The researchers will assess the outcome of LARC use over 12 months by sociodemographic factors (age, race/ethnicity, health insurance), reproductive characteristics (parity, pregnancy intentions, prior contraceptive use) and women's autonomy in contraceptive decision-making including perceptions of bias in education and counseling.
Sub-analyses for unintended pregnancy | 12 months
  The researchers will assess the outcome of unintended pregnancy by sociodemographic factors (age, race/ethnicity, parental education, health insurance, receipt of public assistance) and reproductive characteristics (parity, pregnancy intentions, male partner, prior contraceptive use).
Sub-analyses for certificate or degree completion (ordinal outcome including categories for on-time progression for graduation, delayed progression or dropout), measured by student report (questionnaire) | 12 months
  The researchers will assess the ordinal educational outcome variable by age, race/ethnicity, parental education, and poverty. The researchers will also test interaction of the intervention with race/ethnicity, parental education, and poverty.
Unintended pregnancy incidence | 3 years
  The researchers will measure pregnancy through questionnaires and urine pregnancy tests.
Certificate or degree completion | 3 years
Change in receipt of public assistance (questionnaire) | Baseline, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia C. Harper, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Frost JJ, Lindberg LD, Finer LB. Young adults' contraceptive knowledge, norms and attitudes: associations with risk of unintended pregnancy. Perspect Sex Reprod Health. 2012 Jun;44(2):107-16. doi: 10.1363/4410712. Epub 2012 May 8. PMID 22681426
- [Background] Finer LB, Zolna MR. Shifts in intended and unintended pregnancies in the United States, 2001-2008. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S43-8. doi: 10.2105/AJPH.2013.301416. Epub 2013 Dec 19. PMID 24354819
- [Background] Trieu SL, Bratton S, Hopp Marshak H. Sexual and reproductive health behaviors of California community college students. J Am Coll Health. 2011;59(8):744-50. doi: 10.1080/07448481.2010.540764. PMID 21950256
- [Background] Harper CC, Rocca CH, Thompson KM, Morfesis J, Goodman S, Darney PD, Westhoff CL, Speidel JJ. Reductions in pregnancy rates in the USA with long-acting reversible contraception: a cluster randomised trial. Lancet. 2015 Aug 8;386(9993):562-8. doi: 10.1016/S0140-6736(14)62460-0. Epub 2015 Jun 16. PMID 26091743
- [Background] Sundstrom B, Baker-Whitcomb A, DeMaria AL. A qualitative analysis of long-acting reversible contraception. Matern Child Health J. 2015 Jul;19(7):1507-14. doi: 10.1007/s10995-014-1655-0. PMID 25424456
- [Background] Thompson KM, Rocca CH, Kohn JE, Goodman S, Stern L, Blum M, Speidel JJ, Darney PD, Harper CC. Public Funding for Contraception, Provider Training, and Use of Highly Effective Contraceptives: A Cluster Randomized Trial. Am J Public Health. 2016 Mar;106(3):541-6. doi: 10.2105/AJPH.2015.303001. Epub 2016 Jan 21. PMID 26794168
- [Background] Landry DJ, Wei J, Frost JJ. Public and private providers' involvement in improving their patients' contraceptive use. Contraception. 2008 Jul;78(1):42-51. doi: 10.1016/j.contraception.2008.03.009. Epub 2008 May 29. PMID 18555817
- [Background] Gibbs SE, Rocca CH, Bednarek P, Thompson KMJ, Darney PD, Harper CC. Long-Acting Reversible Contraception Counseling and Use for Older Adolescents and Nulliparous Women. J Adolesc Health. 2016 Dec;59(6):703-709. doi: 10.1016/j.jadohealth.2016.07.018. Epub 2016 Sep 21. PMID 27665153
- [Background] El Ayadi AM, Rocca CH, Kohn JE, Velazquez D, Blum M, Newmann SJ, Harper CC. The impact of an IUD and implant intervention on dual method use among young women: Results from a cluster randomized trial. Prev Med. 2017 Jan;94:1-6. doi: 10.1016/j.ypmed.2016.10.015. Epub 2016 Oct 20. PMID 27773708
- [Background] Rocca CH, Thompson KM, Goodman S, Westhoff CL, Harper CC. Funding policies and postabortion long-acting reversible contraception: results from a cluster randomized trial. Am J Obstet Gynecol. 2016 Jun;214(6):716.e1-8. doi: 10.1016/j.ajog.2015.12.009. Epub 2015 Dec 12. PMID 26692178
- [Background] Harper CC, Henderson JT, Raine TR, Goodman S, Darney PD, Thompson KM, Dehlendorf C, Speidel JJ. Evidence-based IUD practice: family physicians and obstetrician-gynecologists. Fam Med. 2012 Oct;44(9):637-45. PMID 23027156
- [Background] Kost K, Singh S, Vaughan B, Trussell J, Bankole A. Estimates of contraceptive failure from the 2002 National Survey of Family Growth. Contraception. 2008 Jan;77(1):10-21. doi: 10.1016/j.contraception.2007.09.013. Epub 2007 Dec 3. PMID 18082661
- [Background] Rocca CH, Harper CC. Do racial and ethnic differences in contraceptive attitudes and knowledge explain disparities in method use? Perspect Sex Reprod Health. 2012 Sep;44(3):150-8. doi: 10.1363/4415012. Epub 2012 Jun 26. PMID 22958659
- [Background] Finer LB, Zolna MR. Declines in Unintended Pregnancy in the United States, 2008-2011. N Engl J Med. 2016 Mar 3;374(9):843-52. doi: 10.1056/NEJMsa1506575. PMID 26962904
- [Background] Thompson KM, Stern L, Gelt M, Speidel JJ, Harper CC. Counseling for IUDs and implants: are health educators and clinicians on the same page? Perspect Sex Reprod Health. 2013 Dec;45(4):191-5. doi: 10.1363/4519113. Epub 2013 Oct 28. PMID 24325290
- [Background] Harper CC, Stratton L, Raine TR, Thompson K, Henderson JT, Blum M, Postlethwaite D, Speidel JJ. Counseling and provision of long-acting reversible contraception in the US: national survey of nurse practitioners. Prev Med. 2013 Dec;57(6):883-8. doi: 10.1016/j.ypmed.2013.10.005. Epub 2013 Oct 12. PMID 24128950
- [Background] Rocca CH, Goodman S, Grossman D, Cadwallader K, Thompson KMJ, Talmont E, Speidel JJ, Harper CC. Contraception after medication abortion in the United States: results from a cluster randomized trial. Am J Obstet Gynecol. 2018 Jan;218(1):107.e1-107.e8. doi: 10.1016/j.ajog.2017.09.020. Epub 2017 Oct 3. PMID 28986072
- [Background] Kavanaugh ML, Jerman J, Finer LB. Changes in Use of Long-Acting Reversible Contraceptive Methods Among U.S. Women, 2009-2012. Obstet Gynecol. 2015 Nov;126(5):917-927. doi: 10.1097/AOG.0000000000001094. PMID 26444110
- [Background] Moore PJ, Adler NE, Kegeles SM. Adolescents and the contraceptive pill: the impact of beliefs on intentions and use. Obstet Gynecol. 1996 Sep;88(3 Suppl):48S-56S. doi: 10.1016/0029-7844(96)00244-x. PMID 8752228
- [Background] Trussell J. Contraceptive efficacy. In: Hatcher R, Trussell J, Nelson A, Cates W, Kowal D, Policar M, eds. Contraceptive technology, 20th edn. New York: Ardent Media, 2011: 779-863.
- [Background] Whitaker AK, Johnson LM, Harwood B, Chiappetta L, Creinin MD, Gold MA. Adolescent and young adult women's knowledge of and attitudes toward the intrauterine device. Contraception. 2008 Sep;78(3):211-7. doi: 10.1016/j.contraception.2008.04.119. Epub 2008 Jul 3. PMID 18692611
- [Background] Golden SD, Earp JA. Social ecological approaches to individuals and their contexts: twenty years of health education & behavior health promotion interventions. Health Educ Behav. 2012 Jun;39(3):364-72. doi: 10.1177/1090198111418634. Epub 2012 Jan 20. PMID 22267868
- [Background] Foster DG, Biggs MA, Ralph L, Gerdts C, Roberts S, Glymour MM. Socioeconomic Outcomes of Women Who Receive and Women Who Are Denied Wanted Abortions in the United States. Am J Public Health. 2018 Mar;108(3):407-413. doi: 10.2105/AJPH.2017.304247. Epub 2018 Jan 18. PMID 29345993
- [Background] Dehlendorf C, Henderson JT, Vittinghoff E, Steinauer J, Hessler D. Development of a patient-reported measure of the interpersonal quality of family planning care. Contraception. 2018 Jan;97(1):34-40. doi: 10.1016/j.contraception.2017.09.005. Epub 2017 Sep 18. PMID 28935217
- [Derived] Morse SM, Yarger J, Hopkins K, Hecht HK, Rossetto I, Perez LAT, Raymond-Flesch M, Tyler L, Lizarraga M, Hargrave-Bouagnon A, Harper CC. Intimate partner violence and delays in obtaining contraception among young people in California and Texas. Contraception. 2025 Dec;152:111203. doi: 10.1016/j.contraception.2025.111203. Epub 2025 Sep 4. PMID 40914262
- [Derived] Harper CC, Yarger J, Mangurian C, Hopkins K, Rossetto I, Elmes S, Hecht HK, Sanchez A, Hernandez R, Shokat M, Steinberg JR. Mental Health Distress and Delayed Contraception Among Older Adolescents and Young Adults. J Womens Health (Larchmt). 2024 Jul;33(7):870-878. doi: 10.1089/jwh.2023.0549. Epub 2024 Mar 11. PMID 38465503
- [Derived] Yarger J, Hopkins K, Elmes S, Rossetto I, De La Melena S, McCulloch CE, White K, Harper CC. Perceived Access to Contraception via Telemedicine Among Young Adults: Inequities by Food and Housing Insecurity. J Gen Intern Med. 2023 Feb;38(2):302-308. doi: 10.1007/s11606-022-07669-0. Epub 2022 Jun 3. PMID 35657468